CLINICAL TRIAL: NCT01430884
Title: Human Coronary Aspirate: Characterization of Particular and Soluble Substances and the Impact on Microvascular Obstruction
Brief Title: Analysis of Human Coronary Aspirate
Acronym: AHCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Petra Kleinbongard, scientific assistant, Universität Duisburg-Essen
Other Study IDs: ASP-04
Record Dates: First submitted 2011-08-24; First posted 2011-09-08 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Arteriosclerosis; Coronary Heart Disease; No Reflow Phenomenon
Keywords: coronary aspirate blood; particular debris / microemboli; distal occlusion device
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; No-Reflow Phenomenon

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * coronary arterial blood distal to the lesion before stent implantation
  * coronary aspirate blood during stent implantation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aspirate Blood
  Interventions: Other: Aspirated Coronary Blood

INTERVENTIONS:
Other: Aspirated Coronary Blood — Coronary arterial blood is taken distal to the lesion before stent implantation and serve as control and coronary aspirate blood is obtained during stent implantation.

SUMMARY:
During elective percutaneous coronary intervention (PCI), both proximal and distal protection devices are used. The distal occlusion protection device temporarily occludes the vessel distal to the lesion during the intervention, thereby capturing both particular debris and soluble substances released from the lesion such that they can be aspirated and prevented from reaching the coronary microcirculation. Rather than simply discarding the material which is retrieved from use of protection devices, the investigators have recently taken advantage of this situation, sampled the particulate and soluble material and subjected it to a variety of analyses with the ultimate goal to have a better insight into the respective plaque composition and to correlate it to the individual imaging and clinical data. On the basis of such information the investigators aim to better understand the pathophysiology of plaque vulnerability and to possibly predict the clinical development of the individual patient.

DETAILED DESCRIPTION:
Patients

* Symptomatic patients with a significant stenosis (diameter stenosis >75% or significant FFR) in a native coronary vessel or a saphenous vein aortocoronary bypass graft.
* All patients are on aspirin (100 mg/day) and received 10,000 I.U. heparin intravenously.
* Coronary angiography is performed via the femoral approach.
* Full informed consent are obtained from all patients before participating in the study.

Stenosis severity/Plaque composition

* Quantification of stenosis severity was performed with the use of off-line caliper measurements (QCA-MEDIS, Leiden, NL).
* Intravascular imaging analyses before and after stent implantation to characterize plaque morphology:

  1. IVUS(Eagle-EyeTM 20 MHz catheter and R-100 pullback device, Volcano Corporation, Rancho Cordova, CA, USA)
  2. OCT (St. Jude Medical Lightlab C7 Dragonfly Imaging Catheter)
  3. NIRS (InfraReDx TVC Insight catheter)

Interventional procedure

Distal balloon occlusion devices:

* TriAktiv SVG/3.5-FX-catheter; Kensey Nash, Exton, USA or
* GuardWire Temporary Occlusion & Aspiration System; Medtronic Inc., Minneapolis, MN USA Implantation of balloon-expandable stents using balloon pressures between 14 and 18 atm and a balloon-to-vessel diameter ratio of 1:1.

Coronary arterial blood and coronary aspirate

* Coronary arterial blood is taken distal to the lesion before stent implantation and coronary aspirate blood is obtained during stent implantation (each in Heparin- or EDTA- Monovettes, SARSTEDT AG & Co, Nümbrecht, Germany).
* Ex vivo coronary aspirate blood is filtered through a mesh filter with pores of 40 μm diameter.
* Immediately centrifugation of the filtered coronary arterial and aspirate blood (800g, 10 min, 4°C).
* Particulate debris and coronary arterial and aspirate plasma are quickly frozen in liquid nitrogen and stored at -80°C until further use.

Analysis / Aim :

* Using different methods for determining severity of stenosis and plaque composition.
* Using different biochemical methods to characterize particular and soluble substances released during stenting into coronary aspirate.
* Using different bioassays to study vasoconstrictor potential of human coronary aspirate plasma and the impact. of coronary aspirate on the coronary microcirculation and on cardiac contraction.
* Correlation of ex vivo measurements with patients disease and clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with a significant stenosis (diameter stenosis >75% or significant FFR) in a native coronary vessel or a saphenous vein aortocoronary bypass graft

Exclusion Criteria:

* Patients whereby a distal balloon occlusion devices is not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive, symptomatic patients with a significant stenosis in a native coronary vessel or a saphenous vein aortocoronary bypass graft.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2004-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Characterization of particular and soluble substances released during stenting into coronary aspirate and its vasoconstrictor potential. | up to two years
  * biochemical characterization: (quantification (as amount or concentration) of vasoconstrictive substances; cell fragments, proteins and lipids within the aspirate via HPLC, MS, or EIA Kits)
  * in vitro vasoconstriction, coronary microcirculation and cardiac contraction by aspirate (vasoconstriction detected as response of isolated arteries to aspirate normalized to that by KCl in a myograph; coronary microcirculation detected as coronary flow and cardiac contraction as left ventricular pressure within in the in vitro Langendorff heart model)

SECONDARY OUTCOMES:
Correlation of characteristics of soluble and particular substances within aspirate to characteristics of coronary lesion and/or patients underlying disease | up to three years
  e.g.: concentration of vasoconstrictors to plaque composition; concentration of vasoconstrictors to patient underlying disease; amount of particular debris to plaque composition; amount of particular debris to patient underlying disease
Comparison of stenosis severity estimation using QCA and FFR versus IVUS, OCT and NIRS | up to one year
  intra- individual comparison of all parameter for stenosis severity and plaque characterisation

CONTACTS AND LOCATIONS:
Overall Officials: Petra Kleinbongard, PhD, Principal Investigator — Institute of Pathophysiology, University of Essen Medical School
Locations (1):
- Center of Internal Medicine, University of Essen Medical School, Essen, Germany

REFERENCES:
- [Derived] Horn P, Baars T, Kahlert P, Heiss C, Westenfeld R, Kelm M, Erbel R, Heusch G, Kleinbongard P. Release of Intracoronary Microparticles during Stent Implantation into Stable Atherosclerotic Lesions under Protection with an Aspiration Device. PLoS One. 2015 Apr 27;10(4):e0124904. doi: 10.1371/journal.pone.0124904. eCollection 2015. PMID 25915510
- [Derived] Baars T, Konorza T, Kahlert P, Mohlenkamp S, Erbel R, Heusch G, Kleinbongard P. Coronary aspirate TNFalpha reflects saphenous vein bypass graft restenosis risk in diabetic patients. Cardiovasc Diabetol. 2013 Jan 10;12:12. doi: 10.1186/1475-2840-12-12. PMID 23305356